CLINICAL TRIAL: NCT06878079
Title: Assessing Enhanced Recovery After Surgery (ERAS) Intervention Impact on Postoperative Recovery in Gynecological Patients Using QoR-15 Questionnaire
Brief Title: ERAS and Postoperative Recovery in Gynecologic Patients: A QoR-15 Study
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Other Study IDs: 202407159RINB
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Gynecologic; ERAS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERAS care: ERAS emphasizes preoperative education, early interventions (e.g., smoking cessation, anemia management, nutrition optimization), intraoperative strategies (e.g., fluid balance, nausea prevention, temperature control), and postoperative care (e.g., early mobilization, pain control, ileus prevention).
- traditional perioperative care (non-ERAS): Traditional perioperative care (non-ERAS) follows a more conservative approach, often involving prolonged preoperative fasting, liberal fluid administration, routine use of nasogastric tubes, and opioid-based pain management. Postoperatively, patients typically experience delayed oral intake and prolonged bed rest, leading to a longer hospital stay and higher risk of complications such as ileus and deep vein thrombosis.

SUMMARY:
The Quality of Recovery-15 (QoR-15) questionnaire is a widely used Patient-Reported Outcome Measure (PROM) for evaluating postoperative recovery, including pain, physical function, and emotional well-being. Enhanced Recovery After Surgery (ERAS) is a multidisciplinary care model designed to optimize perioperative management through standardized protocols.

For gynecological surgery, ERAS emphasizes preoperative education, early interventions (e.g., smoking cessation, anemia management, nutrition optimization), intraoperative strategies (e.g., fluid balance, nausea prevention, temperature control), and postoperative care (e.g., early mobilization, pain control, ileus prevention). However, while ERAS is gaining acceptance, its effectiveness can vary due to workload, patient variability, and institutional resources, and its superiority over traditional care remains inconclusive.

This study aims to objectively compare ERAS and traditional perioperative care using the QoR-15 questionnaire to assess patient satisfaction, recovery speed, surgical risk reduction, and complication prevention. Rather than solely promoting ERAS, this research seeks to evaluate its applicability, enhance personalized care, and provide scientific evidence for perioperative management optimization.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 80 years.
* Undergoing routine gynecological surgery, including total or subtotal hysterectomy, myomectomy, oophorectomy, gynecologic cancer staging surgery, cytoreductive surgery, and pelvic exenteration.
* Cancer patients with an Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Receiving either standard perioperative care or ERAS protocol-based care.

Exclusion Criteria:

* Age below 20 years.
* Lack of decision-making capacity.
* Undergoing emergency surgery.
* History of clinical depression.
* Undergoing palliative surgery.
* History of chronic pain.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who undergoing routine gynecological surgery, including total or subtotal hysterectomy, myomectomy, oophorectomy, gynecologic cancer staging surgery, cytoreductive surgery, and pelvic exenteration.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery-15 (QoR-15) questionnaire | 5 mins
  The Quality of Recovery-15 (QoR-15) questionnaire is a widely used Patient-Reported Outcome Measure (PROM) for evaluating postoperative recovery, including pain, physical function, and emotional well-being.

IPD SHARING:
Plan to Share IPD: Undecided